CLINICAL TRIAL: NCT06503835
Title: Efficacy of Fluoroscopy Guided Transforaminal Epidural Steroid and Steroid Plus Ozone Injection in Patients With Lumbar Radiculopathy
Brief Title: Efficacy of Transforaminal Epidural Steroid and Its Combination With Ozone in Lumbar Radiculopathy
Status: Completed | Type: Observational
Sponsor: Ibn Sina Hospital (Other Government)
Responsible Party: Principal Investigator, Derya Bayram, Medical Doctor, Pain Specialist, Ibn Sina Hospital
Other Study IDs: IbnSinaH-PM-DB-01
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain; Radiculopathy Lumbar; Hernia; Disk Herniated Lumbar
Keywords: Low back pain; Injections; Steroids; Ozone; Disk Herniated Lumbar
MeSH Terms: conditions — Low Back Pain; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The patients who underwent transforaminal epidural steroid and ozone injection: Patients who received combination therapy were injected 5ml of ozone at a concentration of 28 g/ml and two mL of dexamethasone (8 mg) and 3 mL of saline for each transforaminal epidural injection level under fluoroscopy guidance
  Interventions: Procedure: Fluoroscopy Guided Transforaminal Epidural Ozone Injection; Procedure: Fluoroscopy Guided Transforaminal Epidural Steroid Injection
- The patients who underwent transforaminal epidural steroid injection alone: Patients who received transforaminal epidural steroid injection were injected two mL of dexamethasone (8 mg) and 3 mL of saline for each transforaminal epidural injection level.
  Interventions: Procedure: Fluoroscopy Guided Transforaminal Epidural Steroid Injection

INTERVENTIONS:
Procedure: Fluoroscopy Guided Transforaminal Epidural Ozone Injection — All procedures were performed under light sedation in a sterile operating room. Ozone was created by an ozone generator (Dr. J. Hänsler Ozonosan, Iffezheim, Germany). Appropriate diffusion of the non-ionic contrast agent into the periradicular and epidural area was verified through anteroposterior and lateral fluoroscopic images and the injections were then safely performed. Patients who underwent transforaminal epidural steroid plus ozone injection received additionally 5ml of ozone at a concentration of 28 g/ml for each transforaminal epidural injection level.
  Groups: The patients who underwent transforaminal epidural steroid and ozone injection
Procedure: Fluoroscopy Guided Transforaminal Epidural Steroid Injection — All procedures were performed under light sedation in a sterile operating room.Appropriate diffusion of the non-ionic contrast agent into the periradicular and epidural area was verified through anteroposterior and lateral fluoroscopic images and the injections were then safely performed. Patients who underwent transforaminal epidural steroid injection received two mL of dexamethasone (8 mg) and 3 mL of saline for each transforaminal epidural injection level

SUMMARY:
This retrospective study aimed to assess the clinical effectiveness and safety of transforaminal epidural injections of steroid and ozone mixture versus steroid alone in low back and radicular leg pain related to disk herniation.

DETAILED DESCRIPTION:
Low back and radicular leg pain due to radiculopathy are the common presenting symptoms in the field of pain medicine.For patients with chronic low back and radicular leg pain, pain relief can be achieved through minimally invasive interventional procedures under fluoroscopic guidance. Since some patients may experience persistent pain and the potential development risk of failed back surgery syndrome, minimally invasive procedures are preferred as a pre-surgical intervention.

Interlaminar or transforaminal epidural steroid injections are the most commonly used nonsurgical interventions for disc herniation. Ozone therapy has also started to be used as frequently as steroids. Previous studies have shown that ozone can be given through intradiscally, epidural space, and paravertebral muscles. Ozone gase is thought to modulate levels of cytokines and prostaglandins, minimize reactive oxidant species levels, and improve local periganglionic circulation.

The objective of this study was to assess the short- and long-term clinical efficacy of transforaminal epidural steroid and steroid plus ozone injection in patients presenting with low back and radicular leg pain and to analyze which treatment method is most beneficial in reducing pain relief.

This was a retrospective study of 120 patients who underwent transforaminal epidural steroid or combination of steroid and ozone injection between June and December 2020 in the Ankara University Faculty of Medicine, Department of Pain Medicine.

Demographic information, pain intensity, localization, pattern (neuropathic/nonneuropathic/mix), and patients' quality of life and the treated level (the innervation territories of L2 (Lomber), L3, L4, L5, or S1 (Sacral)) were analyzed. Pain intensity was assessed with the Visual Analog Scale (VAS), and patient disability was evaluated with the Oswestry Disability Questionnaire (ODI).

One group included patients who underwent transforaminal epidural steroid and ozone injection, and another group included patients who underwent transforaminal epidural steroid injection alone. In both groups, two mL of dexamethasone (8 mg) and 3 mL of saline were used for each transforaminal epidural injection level. Patients who received combination therapy were injected 5ml of ozone at a concentration of 28 g/ml in addition to steroids for each level.

The investigators evaluated the patients' records of VAS and ODI scores on the day of the procedure and at the 24th hours (for VAS only) 1st, 3rd, 6th, and 12th months after the procedure. Patients' satisfaction was assessed using modified MacNab scale scores after the 1st and 12th months. The post-treatment results of the patients were compared between the two groups and with the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Files of patients underwent transforaminal epidural steroid or combination of steroid and ozone injection
* Age between 18-75 years
* Body mass index (BMI) <35,
* VAS score ≥ 4
* Radicular pain not responding to conservative therapy related to lumbar disk herniation on magnetic resonance imaging
* Duration of pain of >3 months

Exclusion Criteria:

* Pregnancy
* Major progressive neurologic deﬁcits
* Infective or inﬂammatory diseases
* Uncontrolled diabetes or other severe internal comorbidities
* Malignancy
* international normalized ratio (INR) > 1.2
* Glucose-6-phosphate dehydrogenase deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients (age range, 18-72 years) who underwent transforaminal epidural steroid or combination of steroid and ozone injection between June and December 2020 in the Ankara University Faculty of Medicine, Department of Pain Medicine.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 24th hours, 1st, 3rd, 6th, and 12th months
  The VAS score for pain assessment ranges between 0-10 ( (0=no pain, 5=moderate pain, 10=extremely severe pain).

SECONDARY OUTCOMES:
Oswestry Disability Questionnaire (ODI) | 1st, 3rd, 6th, and 12th months
  ODI is a questionnaire in which the level of disability increases as the total score increases. Total scores vary between 0 and 50.
MacNab Scale Scores | 1st and 12th months
  The MacNab scale scores were used for success in pain decrease and include excellent, good, fair, and poor. The "excellent" and "good" results were accepted as favorable outcomes, and the "fair" and "poor" results were considered unsatisfactory

CONTACTS AND LOCATIONS:
Overall Officials: Derya Bayram, M.D, Principal Investigator — Ankara University Faculty of Medicine, Department of Pain Medicine; İbrahim Aşık, Prof. Dr, Principal Investigator — Ankara University Faculty of Medicine, Department of Pain Medicine
Locations (1):
- Ankara University Faculty of Medicine, İbni Sina Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No